CLINICAL TRIAL: NCT03091335
Title: The Effects of Music Listening on Intra-operative Anxiety in Patients Undergoing Awake Deep Brain Stimulation for Movement Disorders.
Brief Title: Music-listening During Deep Brain Stimulation to Relieve Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Darlene A. Lobel, MD (Other)
Responsible Party: Sponsor-Investigator, Darlene A. Lobel, MD, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-467
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Movement Disorders; Deep Brain Stimulation
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Intervention Model Description: Randomization into two groups: music-listening vs headphones-only
Who Masked: Participant
Masking Description: Participants will be unaware of their randomization group until all pre-operative measures have been acquired.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music-listening group (Experimental): Patients in this group will listen to music of their choosing during the entirety of the awake portion of deep brain stimulation surgery
  Interventions: Other: Music-listening
- Head-phone only group (No Intervention): Patients in this group will receive the same noise-canceling headphones as the patients in the music-listening group. However, they will remain without music per standard of care for awake deep brain stimulation procedures

INTERVENTIONS:
Other: Music-listening — Patients listen to music on headphones
  Arms: Music-listening group

SUMMARY:
This study aims to demonstrate that music listening in patients undergoing awake deep brain stimulation reduces subjective and objective measures of anxiety. Furthermore, the investigators aim to demonstrate that music may alter neuronal firing patterns based on the type of music played and the location in the brain.

DETAILED DESCRIPTION:
While conscious neurosurgical interventions are generally well-tolerated, they often cause some measure of pain and anxiety. Patients have been reported to suffer from recurring distressing recollections of, or dreams about, the surgery and other post-operative, Post-Traumatic Stress Disorder-like sequelae. High anxiety during surgery correlates with post-operative psychological disturbances. Notably, listening to music reduces anxiety in patients undergoing awake surgical procedures. Nonetheless, DBS is typically performed without music because ambient noise typically interferes with interpretation of neuronal recordings. Recording objective and subjective measures of stress during DBS provides a unique opportunity to determine the effect of music on intra-operative patient anxiety levels in patients listening to music compared to non-music listening control patients. The investigators hypothesize that playing music will improve intra-operative anxiety as measured by objective and subjective measures of stress, including blood pressure, heart rate, cortisol levels and anxiety questionnaires. Additionally, previous data in the investigator's lab has demonstrated that the subthalamic nucleus (STN) responds to melodic music by decreasing the average frequency of neuronal firing. The investigator's pilot study also suggests that STN and thalamic neurons respond differently to melodic music; the neurons in the STN increase synchrony of firing, while neurons in the thalamus decrease synchrony of firing over the course of the music clip. The investigators, therefore, aim to characterize the neuronal firing pattern changes in patients undergoing awake DBS procedures in greater detail, drawing from a larger sample size.

ELIGIBILITY:
Inclusion Criteria:

* STN or VIM targeted DBS surgery, awake DBS surgery

Exclusion Criteria:

* No previous DBS surgeries, no history of deafness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Cortisol Response | one year
  Ratio of intra-operative salivary cortisol to pre-operative salivary cortisol in music-listening vs headphones only patients

SECONDARY OUTCOMES:
Blood Pressure | one year
  Changes in blood pressure over time spent awake in surgery in music-listening patients vs headphones only patients
Medication Requirements | one year
  Number and quantity of anti-hypertensives and sedatives required during awake surgery for music-listening vs headphones only patients
Post-operative Recall Questionnaire | one year
  Satisfaction with surgery and subjective experience of whether music or headphones helped anxiety during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Darlene Lobel, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No